CLINICAL TRIAL: NCT05954429
Title: A Study to Explore the Third-line Treatment of Fruquintinib Combined With Serplulimab in Advanced Non-liver-limited Metastatic Colorectal Cancer: a Single-center, Phase 2 Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junjie Peng, Prof., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDCRC87PJJ
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: MSS; serplulimab; fruquintinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab+Fruquintinib (Experimental): Participants will receive serplulimab 300 mg every 3 weeks (Q3W) concurrently with fruquintinib regimen: 5mg (QD) orally for 2 weeks, 1 week off, repeated every 3 weeks. Treatment repeats every 3 weeks until disease progression or intolerable toxicity.
  Interventions: Drug: serplulimab; Drug: Fruquintinib

INTERVENTIONS:
Drug: serplulimab — Serplulimab is an innovative monoclonal antibody targeting PD-1, developed by Shanghai Henlius Biotech, Inc.
  300 mg, q3w Other name: HLX10
Drug: Fruquintinib — 5mg (QD) orally for 2 weeks, 1 week off, repeated every 3 weeks until disease progression or intolerable toxicity.

SUMMARY:
The aim of this clinical trial is to learn about efficacy of fruquintinib combined with serplulimab in patients with microsatellite stabilized mCRC who have failed standard therapy. The main purpose is to explore efficacy, safety and tolerability of the treatment. At the same time, the correlation between biomarkers (including ctDNA, TPS, CPS, tumor mutation burden, lymphocyte subpopulation, cytokines, TCR, intestinal microbes, etc.) and the efficacy and drug resistance mechanism will be analyzed, which could provide reference for determining the advantaged group.

DETAILED DESCRIPTION:
Serplulimab is an anti-PD-1 monoclonal antibody, and fruquintinib is a tyrosine kinase inhibitor that inhibits tumor angiogenesis. Studies have shown that immunotherapy combined with fruquintinib has preliminary efficacy in the treatment of colorectal cancer. Whether serplulimab combined with fruquintinib can improve the prognosis of patients with colorectal cancer remains to be determined. Therefore, the study is to evaluate the efficacy and safety of serplulimab combination with fruquintinib in patients with microsatellite stabilized mCRC who have failed standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, both sexes;
* Patients with histologically or cytologically confirmed unresectable and metastatic CRC
* non-liver-limited metastasis: including no liver metastasis or liver metastasis accompanied by other metastatic lesions, such as lung metastasis, peritoneal metastasis, etc
* Before enrollment, the tumor tissue was pMMR by immunohistochemistry, or MSS or MSI-L by PCR or NGS;
* Have received standard treatment in the past and developed disease progression or intolerance to standard treatment based on RECIST 1.1 during or after standard treatment. Standard treatment should include:

  1. Fluorouracil, oxaliplatin and irinotecan
  2. With or without anti-VEGF monoclonal antibody
  3. For RAS wild-type patients, combined with anti-EGFR monoclonal antibody
  4. For patients with BRAF mutations, BRAF inhibitor therapy is recommended when drugs are available
* Patients with ECOG score of 0-2 and expected survival time ≥3 months, patients who can cooperate to observe adverse reactions and efficacy;
* At least one measurable tumor lesion according to RECIST 1.1 criteria
* Good organ function:

  1. neutrophil ≥1.5*109/L; Platelet ≥100*109/L; Hemoglobin ≥9g/dl; Serum albumin ≥3g/dl;
  2. Thyroid stimulating hormone (TSH) ≤ 1 times the upper limit of normal, T3 and T4 in the normal range;
  3. bilirubin ≤ 1.5 times the upper limit of normal value; ALT and AST≤ 2 times the upper limit of normal;
  4. Serum creatinine ≤ 1.5 times the upper limit of normal, creatinine clearance ≥60ml/min;
  5. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times the upper limit of the normal range, unless the patient is receiving anticoagulant therapy and the PT value is within the intended range for anticoagulant therapy;
  6. Activated partial thromboplastin time (aPTT) ≤ 1.5 times the upper limit of normal;
* There were no serious concomitant diseases that could make the survival time less than 5 years;
* Negative pregnancy test in female subjects (for female patients of childbearing potential); Infertile female patients;
* Male patients of childbearing potential and female patients of childbearing potential and at risk of pregnancy must agree to use adequate contraception for the entire duration of the study and for 12 months after receiving treatment with the protocol;
* Signed and dated informed consent indicating that the patient has been informed about all relevant aspects of the study;
* Patients who are willing and able to comply with the visit schedule, treatment plan, laboratory tests, and other study procedures;
* Willing to comply with the arrangement during the study period can not participate in any other clinical research on drugs and medical devices

Exclusion Criteria:

* Pathological diagnosis of other intestinal tumors, such as gastrointestinal stromal tumor;
* Tumor tissues were dMMR detected by immunohistochemistry, or MSI-H detected by PCR or NGS
* Prior treatment with PD-1 antibody, PD-L1 antibody, or CTLA-4 antibody;
* Previous or concurrent history of other malignant tumors, excluding adequately treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary carcinoma;
* Active autoimmune disease, history of autoimmune disease (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); It does not include autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes on stable doses of insulin; Vitiligo or cured childhood asthma/allergy without any intervention in adulthood;
* A history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation or allogeneic bone marrow transplantation;
* Contraindications to antiangiogenic drugs (such as active bleeding, gastrointestinal bleeding, hemoptysis, etc.);
* History of interstitial lung disease (excluding radiation pneumonitis without steroid treatment) and non-infectious pneumonia;
* Patients with active pulmonary tuberculosis infection detected by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or with a history of active pulmonary tuberculosis infection more than 1 year before enrollment but without regular treatment;
* The subject has active hepatitis B (HBV DNA ≥2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV-RNA above the detection limit of the assay)
* Severe cardiopulmonary and renal dysfunction;
* Have hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
* A history of psychotropic substance abuse, alcohol or drug abuse;
* Other factors that may affect subject safety or trial compliance as judged by the investigator. Severe medical conditions requiring concomitant treatment (including mental illness), serious laboratory abnormalities, or other family or social factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 3 years
  The proportion of participants whose best outcome is complete remission or partial remission

SECONDARY OUTCOMES:
overall survival (OS) | 3 years
  The time between the start of the participants' treatment and their death from any cause
progression-free survival (PFS) | 3 years
  Time from initiation of treatment to disease progression or death from any cause
adverse events | 3 years
  Assessment of the safety profile of regimen according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China